CLINICAL TRIAL: NCT07021521
Title: Efficacy and Safety of Different Doses of Midazolam for 24-Hour Continuous Sedation in Pre-Eclamptic Women Undergoing Cesarean Section
Brief Title: Midazolam Efficacy/Safety in Pre-Eclamptic C-Section Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuji People's Hospital of Zhejiang Province (Other)
Responsible Party: Principal Investigator, Hongmei Xuan, Principal Investigator, Zhuji People's Hospital of Zhejiang Province
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. 2025-0224
Record Dates: First submitted 2025-06-04; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2021-04

CONDITIONS: Midazolam; Pre-eclampsia; Cesarean Section; Efficacy; Safety
MeSH Terms: conditions — Pre-Eclampsia | interventions — Midazolam; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 mg/kg Midazolam (Control Group) (Placebo Comparator): * Received intravenous saline placebo (volume-matched to active doses)
  * Standard epidural anesthesia with 1.6% lidocaine (15-18 mL to T6 level)
  * Hemodynamic monitoring per protocol
  Interventions: Drug: 0 mg/kg Midazolam (Control Group)
- 0.01 mg/kg Midazolam Group (Experimental): * Intravenous midazolam at 0.01 mg/kg (Jiangsu Enhua Pharmaceutical Co., Ltd.)
  * Standard epidural anesthesia as in Arm 1
  * Continuous sedation monitoring for 24 hours post-dose
  Interventions: Drug: 0.01 mg/kg Midazolam Group
- 0.02 mg/kg Midazolam Group (Experimental): * Intravenous midazolam at 0.02 mg/kg
  * Identical anesthesia and monitoring protocols as other arms
  * Primary focus: Dose-response evaluation for sedation efficacy
  Interventions: Drug: 0.02 mg/kg Midazolam Group
- 0.03 mg/kg Midazolam Group (Experimental): * Intravenous midazolam at 0.03 mg/kg (highest tested dose)
  * Enhanced monitoring for hemodynamic effects (MAP, HR, SpO₂)
  * Primary focus: Optimal dose determination balancing efficacy/safety
  Interventions: Drug: 0.03 mg/kg Midazolam Group

INTERVENTIONS:
Drug: 0 mg/kg Midazolam (Control Group) — * Intravenous administration of volume-matched normal saline (0 mg/kg midazolam equivalent)
  * Administered as single bolus prior to epidural anesthesia
  * Served as active comparator for dose-response evaluation
  Arms: 0 mg/kg Midazolam (Control Group)
Drug: 0.01 mg/kg Midazolam Group — * Intravenous midazolam at 0.01 mg/kg (diluted in normal saline)
  * Administered as single bolus over 2 minutes
  * Manufacturer: Jiangsu Enhua Pharmaceutical Co., Ltd. (Approval H19990027)
  Arms: 0.01 mg/kg Midazolam Group
Drug: 0.02 mg/kg Midazolam Group — * Intravenous midazolam at 0.02 mg/kg
  * Identical administration protocol as 0.01 mg/kg group
  * Primary focus: Intermediate dose efficacy/safety assessment
  Arms: 0.02 mg/kg Midazolam Group
Drug: 0.03 mg/kg Midazolam Group — * Intravenous midazolam at 0.03 mg/kg (maximum tested dose)
  * Special hemodynamic monitoring due to dose-dependent MAP effects
  * Primary focus: Optimal dose determination
  Arms: 0.03 mg/kg Midazolam Group

SUMMARY:
This study will compare four different doses of midazolam (0 mg/kg, 0.01 mg/kg, 0.02 mg/kg, and 0.03 mg/kg) administered intravenously to women with pre-eclampsia undergoing cesarean section. The study aims to evaluate how these different doses affect:

The mother's vital signs (oxygen levels, blood pressure, heart rate) The mother's anxiety levels The baby's condition after birth Any potential side effects Participants will be randomly assigned to one of the four dose groups. Medical staff will monitor both mother and baby for 24 hours after the medication is given.

DETAILED DESCRIPTION:
This study aimed to investigate the efficacy and safety of different doses of midazolam for 24-hour continuous sedation in pre-eclamptic women undergoing cesarean section. A total of 124 pre-eclamptic women admitted from April 2021 to April 2023, scheduled for cesarean section at our hospital, were randomly assigned to Group A, Group B, Group C, and Group D, with 31 women in each group. Midazolam was administered intravenously at doses of 0 mg/kg, 0.01 mg/kg, 0.02 mg/kg, and 0.03 mg/kg, respectively. We compared the oxygen saturation (SPO2), mean arterial pressure (MAP), and heart rate (HR) levels before and 30 minutes after drug administration in all four groups. Visual anxiety scores, fetal Kreb's scores, and sedation efficacy indicators (fentanyl dosage, onset time of sedation, mechanical ventilation time) were assessed in the women at 24 hours before and after the surgery. Adverse reactions were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with pre-eclampsia [6] requiring emergency or planned cesarean section
* Age 18-40 years
* No history of midazolam or related drug allergies
* Able to comply with study protocol (no communication barriers)
* No history of mental illness or substance abuse
* Provided informed consent (patient or legal representative)

Exclusion Criteria:

* Concurrent use of drugs interacting with midazolam
* Severe organ dysfunction (heart, liver, or kidneys)
* Participation in other clinical trials potentially affecting results
* Coagulation disorders or hematological conditions
* Inability to adhere to study protocol
* Severe intraoperative complications (e.g., hemorrhage) compromising data reliability
* Additional sedative/analgesic use within 24 hours post-cesarean

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Maternal anxiety reduction using Visual Analog Anxiety Rating Scale (VAS-A) | 24 hours after cesarean section.
  Comparison of anxiety scores using the Visual Analog Anxiety Rating Scale (VAS-A; range 0-10 cm, where 0 = "no anxiety" and 10 = "worst possible anxiety") at 24 hours post-cesarean section among groups receiving different midazolam doses (0, 0.01, 0.02, or 0.03 mg/kg). Higher scores indicate worse anxiety.

SECONDARY OUTCOMES:
Fentanyl consumption during sedation | Intraoperative period through 24 hours post-surgery
  Total fentanyl dosage (μg) required for adequate sedation in each group.
Sedation onset time | 0-60 minutes post-dose
  Time (minutes) from midazolam administration to achieving target sedation level (Ramsay Sedation Scale ≥4).
Mechanical ventilation duration | From surgery completion until extubation (up to 24 hours)
  Total hours of required mechanical ventilation post-cesarean.
Hemodynamic stability (MAP) | 30 minutes post-midazolam administration
  Mean arterial pressure (mmHg) changes from baseline at 30 minutes post-dose.

OTHER OUTCOMES:
Neonatal outcomes by Krebs score | 30 minutes post-midazolam administration
  Krebs score (range 0-12, higher=better) assessing fetal wellbeing at 30 minutes post-drug administration. Components: heart rate, muscle tone, skin color, reflex activity, and respiration.
Adverse event incidence | 0-48 hours post-surgery
  Frequency of hypotension, vomiting, bradycardia, and respiratory depression in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhuji People's Hospital of Zhejiang Province, Shaoxing, Zhejiang, China